CLINICAL TRIAL: NCT04702217
Title: Physical Activity as a Complementary Treatment in Postural Orthostatic Tachycardia Syndrome - Evaluation of a Structured Physical Activity Program in Clinical Practice
Brief Title: Physical Activity as a Complementary Treatment in POTS
Acronym: POTS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has been cancelled due to the pandemic and we are planning on starting a similar study hopefully next year.
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Isabella Kharraziha, MD, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-POTS
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: POTS
Keywords: Exercise; POTS; Training programme; Treatment; Orthostatic intolerance
MeSH Terms: conditions — Motor Activity; Orthostatic Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POTS patients (Experimental): All POTS patients in the study will perform a 16 week-training program. The present study will be using longitudinal comparisons, meaning that the 100 POTS patients are their own controls. The questionnaires and exercise capacity will be compared before and after the 16-weeks training program.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — A 16-week training program consisting of 2-3 visits per week, and 60 minutes per visit. The program will be done as group exercise under supervision from physiotherapists with special interest in POTS.

SUMMARY:
Postural orthostatic tachycardia syndrome (POTS) is a disorder of unknown origin characterized by orthostatic intolerance and increased heart rate (HR) of ≥ 30 beats/minute during orthostasis in the absence of orthostatic hypotension. In addition to the orthostatic intolerance and tachycardia, patients with POTS experience several debilitating symptoms including light-headedness, nausea, blurred vision, fatigue, mental confusion ("brain-fog"), chest pain and gastrointestinal problems. Several potential underlying mechanisms have been suggested for POTS including autonomic denervation, hypovolemia, hyperadrenergic stimulation and autoantibodies against adrenergic receptors. However, none of these proposed mechanisms has yet led to an effective treatment. Physical activity is recommended as a complimentary treatment in POTS in international guidelines. However, less is known regarding how physical activity could successfully be implemented in clinical practice in patients with POTS. Thus, in the current study, we aim to assess the effect of a 16-week specialized physical activity program in POTS.

DETAILED DESCRIPTION:
A total of 100 patients diagnosed with POTS are asked to participate in the study. Prior to start of the training program a special POTS questionnaire (based on the symptoms reported in The BIG POTS Survey), the orthostatic hypotension questionnaire and SF-36 (general health questionnaire) will be completed by the participants. Orthostatic tests are performed during 10 minutes, measuring heart rate and blood pressure after 0, 1, 3, and, if possible, 10 minutes of standing. On a separate occasion, patients will perform a submaximal biking exercise test, while noting symptoms, degree of exertion, achieved effect, pulse and blood pressure reaction. Following this initial evaluation, the training program will be performed during a total time of 16 weeks, which may be non-consecutive but within 6 months in total. The training program consists of 2-3 visits per week, and 60 minutes per visit. The training may be performed on specialized exercise bicycles in supine position or upright position depending on the severity of POTS symptoms. These exercises will be done under the supervision of physiotherapists with special interest in POTS. After the final training session the POTS questionnaire, the orthostatic hypotension questionnaire and SF-36 will be completed once again. In addition, orthostatic tests and submaximal biking exercise test will be performed on a separate occasion soon after the last training session. The present study will be using longitudinal comparisons, meaning that the 100 POTS patients are their own controls. The POTS questionnaire, the orthostatic hypotension questionnaire, SF-36, hemodynamics and exercise capacity will be compared before and after the 16-weeks training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with POTS who have given written informed consent for participation in the study.

Exclusion Criteria:

* Patients with myalgic encephalomyelitis are excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
POTS questionnaire | 6 months
  Subjective symptoms evaluated according to the POTS questionnaire.

SECONDARY OUTCOMES:
Orthostatic hypotension questionnaire | 6 months
  Subjective symptoms evaluated according to the orthostatic hypotension questionnaire.
SF-36 | 6 months
  Evaluation of the SF-36 (general health questionnaire).
Orthostatic tests | 6 months
  Hemodynamic measurements (pulse reaction) during orthostatic testing.
Submaximal biking exercise | 6 months
  Physical capacity measured in watts.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Hamrefors, MD, PhD, Study Director — Department of Clinical Sciences, Malmö, Lund University, Malmö, Sweden and Department of Internal Medicine, Skåne University Hospital, Malmö, Sweden.
Locations (1):
- Skånes Universitetssjukhus Malmö, Department of Cardiology, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winker R, Barth A, Bidmon D, Ponocny I, Weber M, Mayr O, Robertson D, Diedrich A, Maier R, Pilger A, Haber P, Rudiger HW. Endurance exercise training in orthostatic intolerance: a randomized, controlled trial. Hypertension. 2005 Mar;45(3):391-8. doi: 10.1161/01.HYP.0000156540.25707.af. Epub 2005 Feb 7. PMID 15699447
- [Background] Fu Q, Vangundy TB, Galbreath MM, Shibata S, Jain M, Hastings JL, Bhella PS, Levine BD. Cardiac origins of the postural orthostatic tachycardia syndrome. J Am Coll Cardiol. 2010 Jun 22;55(25):2858-68. doi: 10.1016/j.jacc.2010.02.043. PMID 20579544
- [Background] George SA, Bivens TB, Howden EJ, Saleem Y, Galbreath MM, Hendrickson D, Fu Q, Levine BD. The international POTS registry: Evaluating the efficacy of an exercise training intervention in a community setting. Heart Rhythm. 2016 Apr;13(4):943-50. doi: 10.1016/j.hrthm.2015.12.012. Epub 2015 Dec 9. PMID 26690066
- [Background] Shibata S, Fu Q, Bivens TB, Hastings JL, Wang W, Levine BD. Short-term exercise training improves the cardiovascular response to exercise in the postural orthostatic tachycardia syndrome. J Physiol. 2012 Aug 1;590(15):3495-505. doi: 10.1113/jphysiol.2012.233858. Epub 2012 May 28. PMID 22641777
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576